CLINICAL TRIAL: NCT01215084
Title: A Single-Dose, Open-Label, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Oral Fampridine-PR 10 mg in Chinese, Japanese, and Caucasian Adult Healthy Volunteers
Brief Title: A Pharmacokinetics (PK) and Safety Study of Oral Fampridine-PR 10 mg in Chinese, Japanese, and Caucasian Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218HV101
Record Dates: First submitted 2010-09-16; First posted 2010-10-06 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Human Volunteers
MeSH Terms: interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chinese Subpopulation: Fampridine-PR 10 mg (Experimental): Chinese ethnic participants were administered a single dose of Fampridine-PR 10 mgs
  Interventions: Drug: BIIB041 (Fampridine-PR)
- Japanese Subpopulation: Fampridine-PR 10mg (Experimental): Japanese ethnic participants were administered a single dose of Fampridine-PR 10 mgs
  Interventions: Drug: BIIB041 (Fampridine-PR)
- Caucasian Subpopulation: Fampridine-PR 10mg (Experimental): Caucasian ethnic participants were administered a single dose of Fampridine-PR 10 mgs
  Interventions: Drug: BIIB041 (Fampridine-PR)

INTERVENTIONS:
Drug: BIIB041 (Fampridine-PR) — A single 10mg dose tablet by mouth of fampridine prolonged-release (PR) for all participants
  Other Names: AMPYRA®; Dalfampridine; FAMPYRA®

SUMMARY:
The primary objective of the study is to determine the Pharmacokinetic (PK) and safety profiles of fampridine-PR 10 mg in Chinese and Japanese adult healthy volunteers. The secondary objective of this study is to compare the PK and safety profiles of fampridine-PR 10 mg among the Chinese, Japanese, and Caucasian adult healthy volunteers.

DETAILED DESCRIPTION:
The Caucasian group is included to allow comparison of pharmacokinetic and safety data from different race groups to be performed with data obtained from the same study under the same controlled conditions.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Subjects of Chinese or Japanese origin (at least both maternal and paternal grandparents of Chinese or Japanese origin, respectively), or Caucasian subjects. Japanese subjects should be on Japanese diet on a regular basis.
* All male subjects and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 4 weeks after their single dose of study treatment.
* Body Mass Index (BMI) within the range 18.5 to 30 kg/m2 (inclusive).
* Normal urinalysis results as determined by the Investigator for the following parameters: protein, glucose, specific gravity, ketones, urobilinogen, bilirubin, pH, and blood.
* Normal 12-lead ECG as determined by the Investigator.

Key Exclusion Criteria:

* Known history of human immunodeficiency virus (HIV) infection or positive test result for HIV antibodies.
* Known history of hepatitis B or hepatitis C infection, hepatitis B carrier (positive test result for Hepatitis B Surface Antigen [HBsAg]), or hepatitis C infection (positive test result for Hepatitis C virus antibody [HCV Ab]).
* Psychiatric or neurological disorders.
* History of epilepsy or other convulsive disorders.
* Any cardiovascular, renal, gastrointestinal, respiratory, metabolic disorder, or other major disease, as determined by the Investigator.
* Clinically significant abnormal hematology or blood chemistry values at Screening, as determined by the Investigator; or any screening values for alanine aminotransferase (ALT) and aspartate aminotransferase (AST) that are 1.5 times greater than the upper limit of the normal; any clinically significant (as determined by the Investigator) elevated screening values for bilirubin or creatinine; creatinine clearance lower than 80 mL/minute; any low screening values for platelets or hemoglobin; or an out of normal range for white blood cells (WBC).
* History of alcohol abuse (as defined by the Investigator) within the previous 2 years, or a blood screen positive for alcohol.
* History of drug abuse (as defined by the Investigator) within the previous 2 years, or a urine screen positive for cannabinoids, barbiturates, amphetamines, and benzodiazepines.
* Premalignant and malignant disease.
* History of clinically significant severe allergic or anaphylactic reactions.
* Known allergy to pyridine-containing substances.
* Active bacterial or viral infection within the previous month.
* Female subjects who are pregnant or currently breastfeeding.
* Previous participation in another investigational drug study within the last 3 months.
* Treatment with any prescription medication within the 28 days prior to Day -1. (Treatment with pharmaceutical-grade vitamins is allowed provided the dose and regimen have been stable for the 28 days prior to Day -1.)
* Treatment with any over-the-counter products, including herbal-containing and/or caffeine-containing preparations, and/or alternative health preparations and procedures within the 2 days prior to Day -1.
* Donation of blood (500 mL or greater) within 56 days prior to study dosing or plasma donation within 7 days prior to study dosing.
* Inability to comply with study requirements.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events in each ethnic group | Day 1 to Day 7
Observed maximum (peak) plasma 4-aminopyridine (4-AP) concentration (Cmax) | Day 1 (0 to 24 Hours After Dosing)
Time to reach Cmax following study treatment administration (Tmax) | Day 1 (0 to 24 Hours After Dosing)
Area under the time-concentration curve from time zero to infinity (AUC0-∞) | Day 1 (0 to 24 Hours After Dosing)
Apparent elimination half-life (T1/2) | Day 1 (0 to 24 Hours After Dosing)
Renal clearance of the drug from plasma | Day 1 (0 to 24 Hours After Dosing)
Renal clearance as a fraction of total clearance | Day 1 (0 to 24 Hours After Dosing)
Cumulative excreted drug amount at specified sampling intervals (calculated using the concentration data) | Day 1 (0 to 24 Hours After Dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- Research Site, Melbourne, Australia
- Research Site, Shatin, Hong Kong